CLINICAL TRIAL: NCT06896747
Title: Evaluation of the Therapeutic Effects of Mechanically Engineered Umbilical Cord-Derived Stem Cell Exosomes on Endometrial Injury: A Prospective, Non-Randomized, Parallel-Controlled Clinical Study
Brief Title: Evaluating Mechanically Engineered Stem Cell Exosomes for Treating Endometrial Injury: A Clinical Study
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Collaborators: Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, zhangwanlin, Associate Chief Physician, Tang-Du Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024LC2421
Record Dates: First submitted 2025-03-18; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Thin Endometrial Lining; Female Infertility; Intrauterine Adhesions
MeSH Terms: conditions — Infertility, Female; Gynatresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mechanically Engineered Umbilical Cord Mesenchymal Stem Cell-Derived Exosome Group (ME-UCMSC-Exo) (Experimental): Participants in this arm will receive hysteroscopically guided intra-endometrial injection of 1-1.5 mL mechanically engineered umbilical cord mesenchymal stem cell-derived exosomes (ME-UCMSC-Exo) containing approximately 5×10¹⁰ particles/mL during the proliferative phase (Day 3-7 of the menstrual cycle).
  The exosomes are obtained from mechanically preconditioned UC-MSC cultures, which are subjected to biomechanical stress during expansion to enhance regenerative properties.
  The study aims to evaluate the efficacy of ME-UCMSC-Exo in improving endometrial thickness and pregnancy outcomes in patients with thin endometrium secondary to intrauterine adhesions.
  Interventions: Biological: Mechanically Engineered Umbilical Cord Mesenchymal Stem Cell-Derived Exosomes
- Conventional Umbilical Cord Mesenchymal Stem Cell-Derived Exosome Group (UCMSC-Exo) (Experimental): Participants in this arm will receive hysteroscopically guided intra-endometrial injection of 1-1.5 mL conventional umbilical cord mesenchymal stem cell-derived exosomes (UCMSC-Exo) containing approximately 5×10¹⁰ particles/mL during the proliferative phase (Day 3-7 of the menstrual cycle).
  Unlike the ME-UCMSC-Exo group, these exosomes are obtained from standard UC-MSC cultures without mechanical stress preconditioning.
  This group serves as a comparator to determine whether mechanical preconditioning enhances exosome efficacy in endometrial regeneration and pregnancy outcomes.
  Interventions: Biological: Umbilical cord mesenchymal stem cell-derived exosomes
- Platelet-Rich Plasma (PRP) Control Group (Active Comparator): Participants in this arm will receive hysteroscopically guided intra-endometrial injection of 1-1.5 mL autologous PRP following standard PRP preparation protocols during the proliferative phase (Day 3-7 of the menstrual cycle).
  PRP contains growth factors such as platelet-derived growth factor (PDGF), vascular endothelial growth factor (VEGF), and transforming growth factor-beta (TGF-β), which have been shown to improve endometrial receptivity and pregnancy outcomes.
  This group serves as a positive control for assessing the efficacy of exosome-based therapies.
  Interventions: Biological: platelet-rich plasma

INTERVENTIONS:
Biological: Mechanically Engineered Umbilical Cord Mesenchymal Stem Cell-Derived Exosomes — Mechanically engineered umbilical cord mesenchymal stem cell-derived exosomes (ME-UCMSC-Exo) are isolated from umbilical cord-derived mesenchymal stem cells (UCMSCs) subjected to mechanical stress conditioning during in vitro expansion. This process enhances exosome yield, bioactivity, and regenerative capacity. The exosomes are purified via ultracentrifugation and characterized for size, protein markers, and RNA content.
  In this study, ME-UCMSC-Exo is administered via intra-endometrial injection under hysteroscopic guidance. Each participant in this intervention group will receive 1-1.5 mL of exosome solution (containing approximately5*10^10 particles/mL) per injection site during the proliferative phase (Day 3-7 of the menstrual cycle). The aim is to enhance endometrial thickness, receptivity, and pregnancy outcomes in patients with thin endometrium secondary to intrauterine adhesions.
  Other Names: ME-UCMSC-Exo; RH-Exo
  Arms: Mechanically Engineered Umbilical Cord Mesenchymal Stem Cell-Derived Exosome Group (ME-UCMSC-Exo)
Biological: Umbilical cord mesenchymal stem cell-derived exosomes — Umbilical cord mesenchymal stem cell-derived exosomes (UCMSC-Exo) are obtained from standard cultured UCMSCs without mechanical stress preconditioning. These exosomes undergo identical purification and characterization procedures as ME-UCMSC-Exo but lack biomechanical priming. UCMSC-Exo is also administered intra-endometrially via hysteroscopic injection at a dose of 1-1.5 mL (5*10^10 particles/mL) per site.
  Other Names: UCMSC-Exo; TCP-Exo
  Arms: Conventional Umbilical Cord Mesenchymal Stem Cell-Derived Exosome Group (UCMSC-Exo)
Biological: platelet-rich plasma — Platelet-rich plasma (PRP) is an autologous biological preparation obtained from centrifuged whole blood. It contains a high concentration of growth factors, including platelet-derived growth factor (PDGF), transforming growth factor-beta (TGF-β), and vascular endothelial growth factor (VEGF), which promote endometrial regeneration.
  In this study, PRP will be administered via hysteroscopically guided intra-endometrial injection at a dose of 1-1.5 mL per injection site, following standard PRP preparation protocols. This group serves as a positive control for evaluating the efficacy of exosome-based therapies.
  Other Names: PRP
  Arms: Platelet-Rich Plasma (PRP) Control Group

SUMMARY:
The goal of this clinical trial is to evaluate if engineered mechanically umbilical cord-derived stem cell exosomes, or conventional umbilical cord -derived stem cell exosomes, can improve endometrial thickness in women with thin endometrium.

The main questions it aims to answer are:

Can exosomes delivered via subendometrial injection improve endometrial thickness or clinical pregnancy rates compared to PRP (platelet-rich plasma)? Are there significant differences in endometrial thickness between the two treatment groups? Researchers will compare the intervention groups, which one group receives mechanical exosomes and the other receives conventional esosomes via subendometrial injection, to the control group, which receives PRP via the same methods, to see if exosomes provide superior therapeutic effects.

Participants will:

Receive either mechanical exosomesor or conventional esosomes or PRP through subendometrial injection.

Be monitored for changes in endometrial parameters.

DETAILED DESCRIPTION:
This study is a prospective, non-randomized controlled clinical trial designed to evaluate the efficacy and safety of mechanically engineered umbilical cord mesenchymal stem cell-derived exosomes (ME-UCMSC-Exo) and conventional umbilical cord mesenchymal stem cell-derived exosomes (UCMSC-Exo) in the treatment of thin endometrium secondary to severe intrauterine adhesions (IUA) following hysteroscopic adhesiolysis. Thin endometrium is a significant challenge in reproductive medicine, associated with poor embryo implantation rates, recurrent implantation failure (RIF), and increased risk of pregnancy complications. Despite conventional hormonal therapies, effective endometrial regeneration remains a clinical challenge.

Emerging regenerative therapies, including exosome-based interventions, offer promising avenues for enhancing endometrial repair and pregnancy outcomes. Exosomes, extracellular vesicles secreted by stem cells, play a crucial role in tissue regeneration by delivering bioactive molecules such as proteins, microRNAs (miRNAs), and growth factors to target cells. The study aims to determine whether mechanically engineered exosomes, which leverage biophysical modulation during the culture process, demonstrate superior efficacy compared to conventional exosomes and platelet-rich plasma (PRP), a widely used biological intervention for thin endometrium.

Study Design This is a prospective, non-randomized, parallel-controlled study.

Patients will be divided into three groups:

Control Group (PRP Group): Endometrial injection of autologous platelet-rich plasma (PRP).

Conventional Exosome Group: Endometrial injection of UCMSC-derived exosomes. Mechanically Engineered Exosome Group: Endometrial injection of ME-UCMSC-derived exosomes.

Primary endpoint: Change in endometrial thickness. Secondary endpoints: Clinical pregnancy rate, implantation rate, live birth rate, miscarriage rate, and safety assessments (including hypersensitivity reactions, infection, and long-term complications).

Intervention Details Each participant will receive a single intra-endometrial injection using a hysteroscopic-guided 17G needle during the proliferative phase (D3-D7 of the menstrual cycle).

PRP Group: 1-1.5mL PRP per injection site (autologous). UCMSC-Exo Group: 1-1.5mL conventional exosome solution per site. ME-UCMSC-Exo Group: 1-1.5mL mechanically engineered exosome solution per site. Rationale for PRP as a Positive Control PRP is used as a positive control due to its established efficacy in improving endometrial thickness and pregnancy outcomes. Meta-analyses of RCTs have demonstrated that PRP significantly enhances endometrial thickness (MD: 1.23mm, 95% CI: 0.87-1.59, p=0.000) and improves clinical pregnancy rates (RR: 2.04, 95% CI: 1.52-2.76, p=0.000). Additionally, PRP is autologous, safe, and widely used in reproductive medicine, making it a suitable comparative intervention for evaluating the therapeutic efficacy of exosomes.

Eligibility Criteria

Inclusion Criteria:

1. Females aged 20-40 years (inclusive of boundary values);
2. Normal ovarian reserve function (criteria: AFC ≥ 7, AMH > 1.1 ng/mL);
3. History of transcervical resection of adhesions (TCRA);
4. Received PRP treatment after TCRA;
5. At least one embryo transfer (ET) cycle in which they underwent standard ovarian stimulation (fresh cycle) or standard hormone replacement therapy (FET cycle), with an endometrial thickness of <7 mm;
6. Planned to continue IVF/ICSI/FET-assisted conception;
7. Able to accept and adhere to treatment and follow-up and willing to sign an informed consent form.

Exclusion Criteria:

1. Patients with severe systemic diseases, surgical contraindications, or cycle contraindications;
2. Patients with reproductive tract infections, genital tuberculosis, pelvic inflammatory disease, or malignant tumors of reproductive organs;
3. Patients with systemic diseases that cause uterine bleeding;
4. Patients allergic to any drugs, materials, or components used in this study;
5. Patients at high risk for hormone-dependent tumors such as breast cancer or ovarian tumors;
6. Patients with untreated submucosal fibroids of any size (FIGO 0/I/II), uterine fibroids ≥5 cm (FIGO III, IV, V, VI, VII), adenomyosis, unicornuate uterus, bicornuate uterus, or endometrial polyps;
7. Patients with hydrosalpinx ≥3 cm or hydrosalpinx of any size with significant vaginal discharge;
8. Patients with ovarian endometriotic cysts (chocolate cysts) ≥4 cm;
9. Patients who participated in other clinical trials within 3 months before surgery or during the study period;
10. Patients unable to tolerate anesthesia;
11. Patients with genetic abnormalities;
12. Other patients deemed unsuitable for participation in this study by the investigator.

Statistical Considerations & Sample Size Estimated sample size: 90 patients (30 per group). Primary outcome variable: Endometrial thickness increase post-treatment. Sample size calculation based on ANOVA analysis and post-hoc Tukey HSD test to compare all intergroup differences while controlling the familywise error rate at α=0.05.

Considering a 10% dropout rate, a total of 90 patients will be recruited.

Follow-up and Outcome Assessment

Patients will be monitored at multiple time points:

1. Baseline (Pre-intervention assessment).
2. Short-term efficacy evaluations:

   Day of progesterone (P) transformation P+7 days Next embryo transfer cycle (HCG trigger day / FET cycle day of progesterone start).
3. Pregnancy outcomes:

   Biochemical pregnancy (Day 15 post-ET). Clinical pregnancy confirmation (Week 5-6). Live birth rate and perinatal complications (up to 1 year post-intervention).

   Safety evaluations:
4. Immediate adverse reactions (allergic responses, infections).
5. Long-term safety (90-day, 1-year follow-up including tumor markers, liver/kidney function tests, and ultrasound assessments).

Scientific & Clinical Significance This is the first clinical study evaluating mechanically engineered and conventional umbilical cord-derived stem cell exosome therapy for thin endometrium.

If successful, the study will establish a novel, cell-free regenerative therapy for patients with refractory thin endometrium.

Findings could pave the way for future exosome-based treatments in reproductive medicine, expanding therapeutic options for women with uterine factor infertility.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 20-40 years (inclusive of boundary values);
2. Normal ovarian reserve function (criteria: AFC ≥ 7, AMH > 1.1 ng/mL);
3. History of transcervical resection of adhesions (TCRA);
4. Received PRP treatment after TCRA;
5. At least one embryo transfer (ET) cycle in which they underwent standard ovarian stimulation (fresh cycle) or standard hormone replacement therapy (FET cycle), with an endometrial thickness of <7 mm;
6. Planned to continue IVF/ICSI/FET-assisted conception;
7. Able to accept and adhere to treatment and follow-up and willing to sign an informed consent form.

Exclusion Criteria:

1. Patients with severe systemic diseases, surgical contraindications, or cycle contraindications;
2. Patients with reproductive tract infections, genital tuberculosis, pelvic inflammatory disease, or malignant tumors of reproductive organs;
3. Patients with systemic diseases that cause uterine bleeding;
4. Patients allergic to any drugs, materials, or components used in this study;
5. Patients at high risk for hormone-dependent tumors such as breast cancer or ovarian tumors;
6. Patients with untreated submucosal fibroids of any size (FIGO 0/I/II), uterine fibroids ≥5 cm (FIGO III, IV, V, VI, VII), adenomyosis, unicornuate uterus, bicornuate uterus, or endometrial polyps;
7. Patients with hydrosalpinx ≥3 cm or hydrosalpinx of any size with significant vaginal discharge;
8. Patients with ovarian endometriotic cysts (chocolate cysts) ≥4 cm;
9. Patients who participated in other clinical trials within 3 months before surgery or during the study period;
10. Patients unable to tolerate anesthesia;
11. Patients with genetic abnormalities;
12. Other patients deemed unsuitable for participation in this study by the investigator.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2025-06-12 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Endometrial thickness | 30-90days
  The endometrial thickness under ultrasound is measured on the HCG trigger day, oocyte retrieval day, day of progesterone Initiationor or embryo transfer day using transvaginal ultrasound in the sagittal/long-axis plane of the uterus. The measurement is taken at the thickest point within a 1 cm range from the uterine fundus, from the basal membrane on one side, perpendicular across the endometrial cavity line to the basal membrane on the opposite side.

SECONDARY OUTCOMES:
clinical pregnancy | 1-6 months
  A clinical pregnancy is diagnosed based on the presence of ultrasound confirmation of a gestational sac in the uterus.

CONTACTS AND LOCATIONS:
Overall Officials: The Fourth Military Medical University, Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Tang-Du Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Data on primary outcome measures, including endometrial thickness and pregnancy rates, will be shared after study completion. Requests for data access can be made through the corresponding author or institutional repository.
Supporting Information: CSR
Time Frame: Individual participant data will be available upon request starting 6 months after the publication of study results and will remain accessible for 3 years.
Access Criteria: Data access is limited to researchers conducting studies on endometrial regeneration and reproductive medicine. Researchers must submit a proposal detailing their intended data use. Approved applicants will receive access via a secure, password-protected platform under a formal data use agreement (DUA)

REFERENCES:
- [Background] Zhang H, Zhu H, Feng J, Zhang Z, Zhang S, Wang Z, Sun L, Zhang W, Gao B, Zhang Y, Lin M. Reprogramming of Activated Pancreatic Stellate Cells via Mechanical Modulation of Transmembrane Force-sensitive N-cadherin Receptor. J Mol Biol. 2023 Jan 15;435(1):167819. doi: 10.1016/j.jmb.2022.167819. Epub 2022 Sep 8. PMID 36089055
- [Background] Cheng B, Wan W, Huang G, Li Y, Genin GM, Mofrad MRK, Lu TJ, Xu F, Lin M. Nanoscale integrin cluster dynamics controls cellular mechanosensing via FAKY397 phosphorylation. Sci Adv. 2020 Mar 4;6(10):eaax1909. doi: 10.1126/sciadv.aax1909. eCollection 2020 Mar. PMID 32181337
- [Background] Zhang Z, Sha B, Zhao L, Zhang H, Feng J, Zhang C, Sun L, Luo M, Gao B, Guo H, Wang Z, Xu F, Lu TJ, Genin GM, Lin M. Programmable integrin and N-cadherin adhesive interactions modulate mechanosensing of mesenchymal stem cells by cofilin phosphorylation. Nat Commun. 2022 Nov 11;13(1):6854. doi: 10.1038/s41467-022-34424-0. PMID 36369425
- [Background] Zhang C, Zhu H, Ren X, Gao B, Cheng B, Liu S, Sha B, Li Z, Zhang Z, Lv Y, Wang H, Guo H, Lu TJ, Xu F, Genin GM, Lin M. Mechanics-driven nuclear localization of YAP can be reversed by N-cadherin ligation in mesenchymal stem cells. Nat Commun. 2021 Oct 28;12(1):6229. doi: 10.1038/s41467-021-26454-x. PMID 34711824
- [Background] Sun H, Dong J, Fu Z, Lu X, Chen X, Lei H, Xiao X, Chen S, Lu J, Su D, Xiong Y, Fang Z, Mao J, Chen L, Wang X. TSG6-Exo@CS/GP Attenuates Endometrium Fibrosis by Inhibiting Macrophage Activation in a Murine IUA Model. Adv Mater. 2024 May;36(21):e2308921. doi: 10.1002/adma.202308921. Epub 2024 Apr 15. PMID 38588501
- [Background] Zhang W, Tang R, Xiao X, Liu J, Li M, Wang X. A Comparative Study on the Efficacy of Subendometrial Versus Intrauterine Platelet-Rich Plasma Injections for Treating Intrauterine Adhesions: A Retrospective Cohort Study. J Minim Invasive Gynecol. 2025 Apr;32(4):378-385.e1. doi: 10.1016/j.jmig.2024.11.007. Epub 2024 Dec 4. PMID 39643206